CLINICAL TRIAL: NCT05970900
Title: Preoperative Imatinib Mesylate Combined With Rectal-sparing Surgery in Patients With c-KIT Gene-mutant Rectal GIST: an Open-label, Single-arm, Phase III Trial（PIRKER）
Brief Title: Preoperative Imatinib Mesylate Combined With Rectal-sparing Surgery in Patients With c-KIT Gene-mutant Rectal GIST
Acronym: PIRKER
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Fujian Medical University Union Hospital (Other)
Responsible Party: Principal Investigator, 蒋伟忠, Associate professor, Fujian Medical University Union Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2023XHYG0025-01
Record Dates: First submitted 2023-07-23; First posted 2023-08-01 (Actual); Last update posted 2023-08-01 (Actual); Status verified 2023-07

CONDITIONS: Gastrointestinal Stromal Tumor of Rectum
Keywords: Gastrointestinal Stromal Tumor; Rectum; Imatinib mesylate; c-KIT gene; Local resection
MeSH Terms: conditions — Gastrointestinal Stromal Tumors; Piebaldism | interventions — Imatinib Mesylate; Mastectomy, Segmental

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Preoperative Imatinib + local excision (Experimental): Following the attainment of the maximum treatment response through imatinib mesylate administration, typically occurring within 6-12 months, as evidenced by two consecutive imaging evaluations, the tumor exhibited no further reduction in size, thus necessitating the selection of surgical intervention.
  According to the characteristics of the location of the tumor, the surgeon decides the surgical approach based on the existing literature and the availability of surgical equipment, including:
  1. Local transanal resection (TA)
  2. Local resection transsacralapproach
  3. Local resection via perineal approach
  4. Local resection transvaginal approach
  Interventions: Drug: Imatinib Mesylate; Procedure: Local resection

INTERVENTIONS:
Drug: Imatinib Mesylate — 1. For patients with c-KIT exon 11 mutation, imatinib mesylate, 400mg, qd.
  2. For patients with c-KIT exon 9 mutation, imatinib mesylate, 600mg or 800mg, qd.
  Other Names: Gleevec
Procedure: Local resection — According to the characteristics of the location of the tumor, the surgeon decides the surgical approach based on the existing literature and the availability of surgical equipment, including:
  1. Local transanal resection (TA)
  2. Local resection transsacralapproach
  3. Local resection via perineal approach
  4. Local resection transvaginal approach

SUMMARY:
Prior to the implementation of preoperative imatinib mesylate therapy, a considerable percentage (ranging from 34.5% to 67.5%) of individuals diagnosed with rectal gastrointestinal stromal tumors (GIST) underwent abdominoperineal resection (APR), a surgical procedure that involved the removal of the anus and necessitated a permanent colostomy.

This study aims to investigate the safety and viability of an organ-preserving approach involving preoperative imatinib mesylate treatment in conjunction with local resection for rectal GIST, specifically targeting patients with c-KIT gene mutations.

DETAILED DESCRIPTION:
Prior to the implementation of preoperative imatinib mesylate therapy, a considerable percentage (ranging from 34.5% to 67.5%) of individuals diagnosed with rectal gastrointestinal stromal tumors (GIST) underwent abdominoperineal resection (APR), a surgical procedure that involved the removal of the anus and necessitated a permanent colostomy.

Previous studies have established that preoperative administration of imatinib mesylate effectively diminishes the size of rectal gastrointestinal stromal tumors (GIST) and enhances the likelihood of sphincter preservation. After initiating preoperative imatinib mesylate treatment, the sphincter preservation rate has notably escalated from 4.2% to 33.0%-94.9%.

In theory, lymph node resection is not required for Gastrointestinal Stromal Tumors (GIST); the local excision of rectal GIST enables sphincter preservation and yields satisfactory anal function and quality of life (QoL). Various surgical techniques are utilized for local excision, including traditional transanal (TA) and transanal minimally invasive surgery (TAMIS) approaches.

This study aims to explore the safety and feasibility of an organ-preservation strategy of preoperative imatinib mesylate combined with local resection in rectal gastrointestinal stromal tumor (GIST), specifically for patients with c-KIT gene mutations.

ELIGIBILITY:
Inclusion Criteria:

1. Over the age of 18.
2. Newly pathology-diagnosed rectal GIST
3. Tumor > 2cm; local resection of R0 is not possible in the initial evaluation.
4. The lower margin of the tumor is ≤ 5cm from the anal verge.
5. C-KIT gene mutation.
6. Male or non-pregnant female.
7. ECOG score 0-2.
8. Did not receive targeted therapy before the start of the clinical trial.
9. Sufficient organ functions are defined as follows:

   Total bilirubin < 1.5×ULN (upper limit of normal, ULN), serum AST (SGOT) and ALT (SGPT) < 2. 5 × ULN, creatinine < 1.5×ULN, neutrophil count > 1. 5 ×109 / L, platelet > 100 × 109 / L.
10. The patient's informed consent has been obtained.

Exclusion Criteria:

1. Pathology is non-rectal GIST.
2. Under the age of 18.
3. Patients with distant metastasis.
4. The patient is not permitted to have additional primary malignant tumors within five years unless those tumors are currently deemed clinically insignificant and do not necessitate active intervention, such as basal cell skin cancer or cervical cancer in situ. The presence of any other malignant diseases is strictly prohibited.
5. Individuals diagnosed with stage III or IV cardiac conditions, specifically congestive heart failure and myocardial infarction occurring within six months prior to the commencement of the study.
6. The patient presents with severe and/or uncontrolled medical ailments, such as unmanaged diabetes, advanced chronic kidney disease, or active uncontrolled infection.
7. Co-administration of imatinib with warfarin or acetaminophen is contraindicated, necessitating the substitution of alternative medications (e.g., low molecular weight heparin in place of warfarin).
8. Subjects undergoing radiotherapy, chemotherapy, and/or targeted therapy.
9. Pregnant or lactating female patients.
10. Cognitive or psychiatric disorders.
11. Profound cardiac, hepatic, and renal dysfunction.
12. Non-adherence by the patient or the researchers' assessment of the patient's inability to complete the entire trial.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Estimated)
Dates: Start 2023-10-01 (Estimated); Primary Completion 2026-10-01 (Estimated); Study Completion 2029-10-01 (Estimated)

PRIMARY OUTCOMES:
Organ preservation | 18 months
  Rectum intact, owing to no total mesorectal excision (TME), no locoregional regrowth unless amenable to limited, curative (R0) salvage surgery by local excision (LE) and no permanent stoma (including a never reversed protective stoma, or a stoma owing to toxicities and/or poor functional outcomes)

SECONDARY OUTCOMES:
3-year disease-free survival | 36 months
  The proportion of participants who remain disease-free at 3 years after surgery
Local recurrence rate | 36 months
  The local recurrence rate is defined as the incidence detection of a tumor involving the bowel wall only that occurs after LE or TME
Overall survival | 36 months
  The proportion of participants who remain survival at 3 years after surgery
R0 resection rate | 18 months
  The R0 resection rate is defined as the rate of R0 resection
Quality of life based on EORTC-QLQs-C30 and EORTC-QLQs-CR29 | Baseline, 3 months, 12 months, 24 months, and 36 months after surgery
  Quality of life accessed by EORTC-QLQs-C30 and EORTC-QLQs-CR29 questionnaire
Anorectal function | Baseline, 3 months, 12 months, 24 months, and 36 months after surgery
  Anorectal function based on LARS score

CONTACTS AND LOCATIONS:
Overall Officials: Weizhong Jiang, MD, Principal Investigator — Fujian Medical University Union Hospital
Locations (1):
- Weizhong Jiang, Fuzhou, Fujian, China

IPD SHARING:
Plan to Share IPD: No